CLINICAL TRIAL: NCT07010692
Title: Using Fractional Lasers and Tirbanibulin Ointment to Treat Keratinocyte Carcinomas
Brief Title: Treating Basal and Squamous Cell Carcinomas With Fractional Laser and Tirbanibulin Ointment
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bruce Robinson, MD (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 25-06-003-2015
Record Dates: First submitted 2025-05-30; First posted 2025-06-08 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Keratinocyte Carcinoma; Basal Cell Carcinomas; Squamous Cell Carcinoma; Skin Cancer
Keywords: Basal Cell Carcinoma; Squamous Cell Carcinoma; BCC; SCC; keratinocyte carcinoma; skin cancer; laser treatment
MeSH Terms: conditions — Carcinoma, Basal Cell; Carcinoma, Squamous Cell; Skin Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Fractional Laser Only (Active Comparator): Treatment of superficial or in situ carcinomas will be with fractional laser only.
  Interventions: Device: non-ablative fractional laser
- Fractional Laser and Tirbanibulin Ointment (Active Comparator): Treatment of nodular or invasive carcinomas will be with fractional laser followed by a course of Klisyri ointment.
  Interventions: Drug: Tirbanibulin ointment 1%; Device: non-ablative fractional laser

INTERVENTIONS:
Drug: Tirbanibulin ointment 1% — Tirbanibulin ointment is applied for 5 nights following the in-office fractional laser procedure for patients with more advanced carcinomas.
  Arms: Fractional Laser and Tirbanibulin Ointment
Device: non-ablative fractional laser — Every skin cancer will be treated with two wavelengths (1550nm and 1927nm) of a non-ablative fractional laser.

SUMMARY:
The investigators seek to evaluate the effectiveness of fractional laser therapy and tirbanibulin ointment to treat squamous and basal cell carcinomas. This will be executed by using both thulium and erbium lasers on previously biopsy-confirmed SCCs and BCCs and applying bulk heating methods. Then, depending on the level of invasiveness, subjects may be instructed to apply the ointment over the course of five nights immediately following the treatment. The intention of this study is to minimize the need for invasive surgical procedures so as to optimize the cosmetic appearance, and provide a treatment option that is beneficial for a wide range of individuals.

ELIGIBILITY:
Inclusion Criteria: biopsy confirmed squamous and/or basal cell carcinoma not previously treated by another method.

Exclusion Criteria:

* Cannot be pregnant at the time of treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-05-16 (Actual); Primary Completion 2030-05 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
Clearance of skin cancer by evidence of no clinical and/or histological recurrence after 5 years. | From enrollment to the end of follow-up monitoring at 5 years.
  Participants will be monitored at 1 month post-procedure then biannually thereafter for 5 years. Site with be observed for clinical recurrence. Optional biopsy at each visit.

SECONDARY OUTCOMES:
Recurrence rate/Appearance/Patient Satisfaction as compared to accepted alternatives (Surgical excision, Mohs, Electrodesiccation and curettage) | Ongoing review from enrollment to the end of 5 year follow-up period & also a final review at the end of 5 years for all participants.
  Review the overall success of the treatment (recurrence and failure rates, appearance, patient satisfaction) compared to traditionally accepted alternative treatments including surgical excision, Mohs surgery, and Electrodesiccation and curettage

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Robinson, MD, Principal Investigator — Bruce Robinson, MD
Locations (1):
- Bruce Robinson, MD, New York, New York, United States

REFERENCES:
- [Result] Robinson BP, Nanni GM. Utilizing fractional lasers and tirbanibulin ointment to treat squamous and basal cell carcinomas. Arch Dermatol Res. 2024 Oct 14;316(10):683. doi: 10.1007/s00403-024-03423-0. PMID 39400600
- See also: Related Info — https://www.brucerobinsonmd.com

DOCUMENTS (1):
  • Study Protocol (2025-05-16): https://cdn.clinicaltrials.gov/large-docs/92/NCT07010692/Prot_000.pdf